CLINICAL TRIAL: NCT01106261
Title: A Randomised Trial of Pulmonary Metastasectomy in Colorectal Cancer
Acronym: PulMiCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); University of Cambridge (Other); University of Sussex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Reference No: 08/0390; CRUK/09/022 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2010-04-13; First posted 2010-04-19 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Pulmonary Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metastasectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulmonary metastasectomy (Experimental): Pulmonary metastasectomy
  Interventions: Procedure: Metastasectomy
- Active monitoring (Active Comparator): Active monitoring
  Interventions: Procedure: Active monitoring

INTERVENTIONS:
Procedure: Metastasectomy — Pulmonary Metastasectomy
  Arms: Pulmonary metastasectomy
Procedure: Active monitoring — Active monitoring
  Arms: Active monitoring

SUMMARY:
Patients who have been treated successfully for bowel cancer (colorectal cancer) sometimes go on to develop nodules of disease in another part of the body. If this disease is found to be related to the original cancer it is called a metastasis. Some patients develop one or more metastases particularly in the lungs or the liver.

There is a growing trend to remove lung metastases with an operation, in the belief that this will help patients live longer, however there have not been any scientific studies to prove this. There is also very little published information about the side effects of this surgery and how it affects subsequent daily living. This is a feasibility study to determine whether it will be possible to conduct a large randomised controlled trial investigating the value of pulmonary metastasectomy (surgery to remove lung metastases) in patients who have been successfully treated for colorectal cancer. There is a two stage consent and randomisation process. Firstly, patients will be invited to consent to having a full range of investigations to assess their suitability for surgery. If found to be suitable, they will then be invited to consent to randomisation between active monitoring of their disease or active monitoring with pulmonary metastasectomy. Patients will be followed up regularly for 5 years to assess their disease status and to measure their quality of life and lung function.

DETAILED DESCRIPTION:
Colorectal cancer is one of the three commonest solid tumours. Approximately 100 cases are diagnosed each day in the UK. In 2006, 37,514 cases of colorectal cancer were diagnosed.

The increasing use of CT scans in routine follow up of patients has led to earlier diagnosis of isolated and/or subclinical lung nodules and there has been widespread adoption of pulmonary metastasectomy in selected cases. A survey of practice in Europe showed that pulmonary metastasectomy is very commonly performed but criteria vary widely. About 300 such operations were being carried out annually in the UK when PulMiCC opened as a 'feasibility' study.

Although well-established in clinical practice there have been no previous randomised controlled trials of the effect of lung metastasectomy on survival and there is doubt as to its clinical effectiveness. The most recent systematic review and meta-analysis concludes that pulmonary metastasectomy is associated with a high likelihood of recurrence, with doubling of the recurrence rate with each of three adverse prognostic factors: (i) more than one metastasis, (ii) an interoperative interval (primary resection to lung metastasectomy) less than three years, (iii) elevated CEA.

In a prospective registry capturing more than 60% of Spanish practice for a two year period these limits were commonly exceeded.

In an RCT it has been shown that recurrence can be detected earlier with CT and/or CEA surveillance and as a result more liver and lung metastasectomy operations were performed. However, these operations did not provide any survival benefit, within the RCT. The uncertainty about the practice has been set out in the British Medical Journal in 2014.

Pulmonary metastasectomy is thus part of a bigger question about effectiveness of surgery for metastases from colorectal cancer.

There are known unfavourable prognostic factors which include the number of metastases and the length of time they take to become evident radiologically: (a) a solitary nodule appearing after a long interval is will be removed in most instances, (b) surgery is rarely advocated when there are multiple metastases present at the time of surgery on the primary colorectal cancer or appearing soon after.

These scenarios represent opposite ends of the continuum of favourable to adverse factors for survival after resection of pulmonary metastases. Most patients operated on fall between these extremes and it is evident that if there is a "yes" towards one end of the continuum and "no" towards the other that there must be cross over zone where there is clinical uncertainty. PulMiCC aims to investigate the outcome following pulmonary metastasectomy in patients where there is accepted clinical uncertainty, to provide evidence to guide practice in the future.

It has also been shown previously that trials requiring patients to consider randomisation between treatments that appear very different, as in this instance between surgery or no surgery, can experience recruitment difficulties. This is because potential participants may have acquired a strong preference for one of the treatments over the other and they are not willing to accept the possibility of being allocated to the less non-preferred option alternative.

There can also be problems of bias if one treatment is mentioned to the patient before the option of a trial is introduced; the first mentioned treatment may be perceived to be preferred between doctor and patient. This trial has been designed to overcome these potential difficulties and maximise recruitment as follows.

Colorectal cancer patients presenting with pulmonary metastases will first be consented for registration into the study. This consent is to undergo evaluation according to the trial protocol as part of the work up for consideration by the MDT. Following evaluation, the MDT will consider how they would normally treat each patient according to their standard local practice. Patients eligible for randomisation will be those for whom clinical uncertainty exists as to whether surgery would be of benefit. This trial design was successful in a study of the feasibility of randomising patients in a trial of mesothelioma surgery.

The time taken for patients to undergo the full range of tests for evaluation gives them time to think carefully about the possible treatment options and discuss them with their doctor. In addition to the patient information leaflet, patients will be invited to take home a DVD explaining the trial in detail, which can be watched as often as the patient likes. It is hoped that those who are ultimately identified as eligible for randomisation will have fewer anxieties because of their extended opportunity to consider the trial.

Local site research staff involved in recruiting patients will attend a training session to learn the best method of informing patients about the trial before recruitment commences.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary colorectal cancer who have undergone resection of the primary cancer with intent to cure, local control has been confirmed and no clinical indications of other active colorectal cancer other than the known lung metastases.

Exclusion Criteria:

* Previous malignancy likely to interfere with protocol treatment or measurement of endpoints, any concurrent illness which could interfere with the treatment protocol or confound survival, unavailable for follow up and assessment according to protocol, psychiatric or mental incapacity that precludes fully informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-12-02 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | 2 years
  We wish to measure the monthly recruitment rate from approximately 11-12 centres over 2 years. This feasibility study aims to determine whether it will be possible to recruit sufficient patients to conduct a larger randomised trial which would be powered to measure survival as the primary outcome.

SECONDARY OUTCOMES:
Survival | 5 years
  Overall survival, Relapse free survival, Lung function (measured by FEV1), Patient reported quality of life (STAI, FACT-An-L and EQ-5D questionnaires), Health economic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Tom Treasure, MD, MS, FRCS, Principal Investigator — UCL
Locations (24):
- Henan Cancer Hospital/The affiliated Cancer Hospital, Zhengzhou, China
- Policlinico Hospital, Catania, Italy
- Institute for Lung diseases of Vojvodina, Kamenitz, Serbia
- United Kingdom (21):
  - Basildon University Hospital, Basildon
  - Birmingham Heartlands Hospital, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Queen's Hospital, Burton-on-Trent
  - Velindre Cancer Centre, Cardiff
  - Golden Jubilee National Hospital, Glasgow
  - Glenfield Hospital, Leicester
  - Liverpool Heart & Chest Hospital, Liverpool
  - The Whittington Hospital, London
  - Royal Free Hospital, London
  - Guy's and St Thomas' NHS Trust, London
  - St George's Hospital, London
  - Royal Brompton Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Papworth Hospital NHS Trust, Papworth Everard
  - Derriford Hospital, Plymouth
  - Sheffield Teaching Hospitals, Sheffield
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Result] Milosevic M, Edwards J, Tsang D, Dunning J, Shackcloth M, Batchelor T, Coonar A, Hasan J, Davidson B, Marchbank A, Grumett S, Williams NR, Macbeth F, Farewell V, Treasure T. Pulmonary Metastasectomy in Colorectal Cancer: updated analysis of 93 randomized patients - control survival is much better than previously assumed. Colorectal Dis. 2020 Oct;22(10):1314-1324. doi: 10.1111/codi.15113. Epub 2020 Jun 14. PMID 32388895
- [Derived] Treasure T, Farewell V, Macbeth F, Batchelor T, Milosevic M, King J, Zheng Y, Leonard P, Williams NR, Brew-Graves C, Morris E, Fallowfield L; PulMiCC investigators. The Pulmonary Metastasectomy in Colorectal Cancer (PulMiCC) burden of care study: Analysis of local treatments for lung metastases and systemic chemotherapy in 220 patients in the PulMiCC cohort. Colorectal Dis. 2021 Nov;23(11):2911-2922. doi: 10.1111/codi.15833. Epub 2021 Aug 2. PMID 34310835
- [Derived] Treasure T, Farewell V, Macbeth F, Monson K, Williams NR, Brew-Graves C, Lees B, Grigg O, Fallowfield L; PulMiCC Trial Group. Pulmonary Metastasectomy versus Continued Active Monitoring in Colorectal Cancer (PulMiCC): a multicentre randomised clinical trial. Trials. 2019 Dec 12;20(1):718. doi: 10.1186/s13063-019-3837-y. PMID 31831062